CLINICAL TRIAL: NCT01209741
Title: An Open Label, Randomized, 3-Period Crossover Study to Evaluate the Comparative Bioavailability of Variably Aged MK-0974 Capsules Administered Orally as Single Doses in Healthy Male and Female Subjects
Brief Title: Bioavailability of Variably Aged MK-0974 Tablets (MK-0974-038)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0974-038
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

ARMS (3):
- 1 (Active Comparator): MK-0974 12MoRT
  Interventions: Drug: telcagepant potassium
- 2 (Active Comparator): MK-0974 5Mo5C
  Interventions: Drug: MK-0974 5Mo5C
- 3 (Active Comparator): MK-0974 12Mo5C
  Interventions: Drug: MK-0974 12Mo5C

INTERVENTIONS:
Drug: telcagepant potassium — [INTERVENTION NAME: MK-0974 12MoRT] Single dose MK-0974 12MoRT (12 month aged MK-0974 capsules, stored at room temperature) 300 mg in one of three treatment periods
  Arms: 1
Drug: MK-0974 5Mo5C — Single dose MK-0974 5Mo5C (5 month aged MK-0974 capsules, stored at 5 Â°C) 300 mg in one of three treatment periods
  Arms: 2
Drug: MK-0974 12Mo5C — Single dose MK-0974 12Mo5C (12 month aged MK-0974 capsules, stored at 5 Â°C) 300 mg in one of three treatment periods
  Arms: 3

SUMMARY:
This study will evaluate the comparative bioavailability of three capsule formulations of MK-0974.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject is a nonsmoker
* Subject is willing to comply with the study restrictions

Exclusion Criteria:

* Subject has a history of stroke, chronic seizures, or major neurological disorder
* Subject has a history of cancer
* Subject is a nursing mother
* Subject has or has a history of any illness that might make participation in the study unsafe or confound the results of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC(0 to infinity) following single dose administration of MK-0974 12Mo5C and 5Mo5C formulations | Through 48 hours postdose
Peak plasma concentration (Cmax) following single dose administration of MK-0974 12Mo5C and 5Mo5C formulations | Through 48 hours postdose

SECONDARY OUTCOMES:
Area under the curve (AUC(0 to infinity) following single dose administration of MK-0974 12MoRT and 5Mo5C formulations | Through 48 hours postdose
Peak plasma concentration (Cmax) following single dose administration of MK-0974 12MoRT and 5Mo5C formulations | Through 48 hours postdose